CLINICAL TRIAL: NCT02428582
Title: Covered Stents Versus Bare-Metal Stents in Chronic Atherosclerotic Gastrointestinal Ischemia
Brief Title: Covered Stents Versus Bare-Metal Stents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Trialbureau radiology, Coordinating trialbureau, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MEC-2013-476
Record Dates: First submitted 2015-04-15; First posted 2015-04-29 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Gastrointestinal Vascular Conditions; Arteriosclerosis; Lifestyle-related Condition; Stenosis; Vascular Insufficiency; Necrosis
Keywords: endovascular treatment; arterial occlusive disease; bare metal stent; polytetrafluoroethylene covered stent
MeSH Terms: conditions — Arteriosclerosis; Mental Disorders; Constriction, Pathologic; Necrosis; Arterial Occlusive Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- bare stent inserted (Active Comparator): Standard bare stent will be placed
  Interventions: Device: Bare stent (Brand Cordis Type Palmaz Blue)
- Covered stent inserted (Experimental): Covered stent will be placed
  Interventions: Device: Covered stent (Atrium Type V12)

INTERVENTIONS:
Device: Covered stent (Atrium Type V12) — An endovascular treatment that consists of inserting a covered stent into the stenosed vessels.
  Arms: Covered stent inserted
Device: Bare stent (Brand Cordis Type Palmaz Blue) — An endovascular treatment that consists of inserting a stent into the stenosed vessels.
  Other Names: Brand Cordis Type Palmaz Blue
  Arms: bare stent inserted

SUMMARY:
To compare the outcome of revascularisation the gastrointestinal arteries using covered stents compared to bare-metal stents in patients with CGI.

DETAILED DESCRIPTION:
Symptomatic chronic atherosclerotic gastrointestinal ischemia (CGI) is an uncommon, potentially underdiagnosed condition caused by fixed stenosis or occlusion of in most conditions at least one of the three gastrointestinal arteries. Atherosclerosis is a predisposing factor for CGI. Clinical symptoms can vary widely. Typical symptoms are postprandial abdominal pain, unintended weight loss and food avoidance. But atypical abdominal pain such as exercise related pain, diarrhoea and nausea can also indicate CGI. The use of endovascular techniques for revascularization of chronic stenosis and occlusions of the gastrointestinal arteries has rapidly increased and endovascular therapy with stenting has become the most common method chosen for revascularization, having replaced open surgery with its associated morbidity and mortality. Nowadays standard care in significant chronic gastrointestinal ischemia is the use of bare metal stents although the patency of these stents is not very high. According retrospective data the patency of covered stents is significantly higher compared to bare metal stents. One likely explanation for these lower restenosis and re-intervention rates observed with covered stents is the established barrier to tissue ingrowth. Only recent retrospective data about this topic is available but the expectancy in this prospective study is that the patency of covered stents is indeed higher compared to metal stents.

ELIGIBILITY:
Inclusion Criteria:

* Patients with consensus diagnostic of CGI based on a clinical meeting with a gastroenterologist, a vascular surgeon and an interventional radiologist.
* Diagnostic consensus of CGI is based on.
* Presence of postprandial pain
* Unexplained weight loss (>5% of normal body weight).
* Significant stenosis of >50% of at least one of the gastrointestinal arteries on a recent CTA (Computer Tomographic Angiography) not older than one year, with maximum slice thickness 1 mm and enhancement in aorta of 300HU (Hounsfields Units)
* Mucosal ischemia detected by VLS (Visible Light Spectroscopy) or tonometry
* Patients over the age of 18 years.
* Patients who gave informed consent.
* Patients have sustained atherosclerosis.

Exclusion Criteria:

* Patients who don't give informed consent.
* Age < 18 years
* No stenosis detected during arteriography.
* Renal insufficiency (GFR below 30 ml/min or GFR below 60 ml/min when comorbidities relevant to kidney function present).
* Previous stent placement in the to be treated gastrointestinal artery.
* Pregnancy
* Celiac artery compression syndrome.
* Vasculitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2016-05; Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
The difference of primary and secondary patency rates of covered stents versus bare-metal stents to treat atherosclerotic CGI disease. | 12 to 24 months

SECONDARY OUTCOMES:
The freedom from restenosis after 6-, 12- and 24- months after stent implantation | 6 to 24 month
  Restenosis is defined as >50% intra-stent stenosis regardless of whether the patient has clinical symptoms
The freedom from symptom recurrence after 6-, 12- and 24- months after stent implantation | 6 to 24 month
  Symptom recurrence is defined as occurrence of clinical symptoms typical for CGI regardless of stent patency
The freedom from reintervention after 6-, 12- and 24- months after stent implantation | 6 to 24 month
  Re-intervention is defined as intervention due to symptom occurrence in the presence of >50% intra -stenosis, either a reimplantation of stent or a surgical procedure.
The clinical outcome in terms of quality of life and therapeutic and total costs after 6-, 12- and 24- months after stent implantation | 6 to 24 month
The clinical outcome in terms therapeutic and total costs after 6-, 12- and 24- months after stent implantation | 6 to 24 month

CONTACTS AND LOCATIONS:
Overall Officials: Adriaan Moelker, dr, Principal Investigator — Erasmus Medical Center
Locations (1):
- ErasmusMC, Rotterdam, South Holland, Netherlands

REFERENCES:
- [Derived] Terlouw LG, van Dijk LJD, van Noord D, Bakker OJ, Bijdevaate DC, Erler NS, Fioole B, Harki J, van den Heuvel DAF, Hinnen JW, Kolkman JJ, Nikkessen S, van Petersen AS, Smits HFM, Verhagen HJM, de Vries AC, de Vries JPM, Vroegindeweij D, Geelkerken RH, Bruno MJ, Moelker A; Dutch Mesenteric Ischemia Study Group. Covered versus bare-metal stenting of the mesenteric arteries in patients with chronic mesenteric ischaemia (CoBaGI): a multicentre, patient-blinded and investigator-blinded, randomised controlled trial. Lancet Gastroenterol Hepatol. 2024 Apr;9(4):299-309. doi: 10.1016/S2468-1253(23)00402-8. Epub 2024 Jan 29. PMID 38301673
- [Derived] van Dijk LJD, Harki J, van Noord D, Verhagen HJM, Kolkman JJ, Geelkerken RH, Bruno MJ, Moelker A; Dutch Mesenteric Ischemia Study group (DMIS). Covered stents versus Bare-metal stents in chronic atherosclerotic Gastrointestinal Ischemia (CoBaGI): study protocol for a randomized controlled trial. Trials. 2019 Aug 20;20(1):519. doi: 10.1186/s13063-019-3609-8. PMID 31429792